CLINICAL TRIAL: NCT05922657
Title: A Prospective, Observational, Multi-center Study to Gather Real World Use Data on the Effectiveness, Safety, and Site-of-service of the Cerene Device
Brief Title: A Registry to Gather Real World Use Data on the Cerene® Cryotherapy Device
Acronym: Progress
Status: Recruiting | Type: Observational
Sponsor: Channel Medsystems (Industry)
Responsible Party: Sponsor
Other Study IDs: PTL-2023-N01
Record Dates: First submitted 2023-06-12; First posted 2023-06-28 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Heavy Menstrual Bleeding; Abnormal Uterine Bleeding; Menorrhagia
Keywords: Cerene; Registry; Cryoablation
MeSH Terms: conditions — Menorrhagia; Metrorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treated patients: This is a registry study with no active intervention outside standard of care. Women will be treated with Cerene per standard of care.
  Interventions: Device: Cerene

INTERVENTIONS:
Device: Cerene — Real world use of Cerene.

SUMMARY:
Channel Medsystems, Inc., the manufacturer of the Cerene® Cryotherapy Device (Cerene), is initiating a prospective, observational registry, the Progress registry, to gather data during real world utilization of the Cerene® Cryotherapy Device (Cerene). The primary objective of this registry is to bridge the gap between clinical results and outcomes achieved and reported during the pivotal study of Cerene and those obtained during its real-world use.

DETAILED DESCRIPTION:
Cerene was approved by the FDA in March 2019 for endometrial cryoablation in premenopausal women with heavy menstrual bleeding due to benign causes for whom child bearing is complete. The primary objective of the Progress registry is to bridge the gap between clinical results and outcomes reported during the pivotal study of Cerene (the CLARITY Study) and those observed during its real-world use. The Progress registry will gather prospective, observational data on up to 300 women that underwent a Cerene treatment. Patients and physicians will complete surveys. Surveys will include patient demographic characteristics and quality of life measures at baseline, procedural details, and post-operative clinical outcomes and quality of life measures.

Patient participation is expected to last approximately 13 months, from the time of patient enrollment to 12 months post treatment. The study will end after the last participating patient in completes her 12 month visit.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for a Cerene treatment
* 25 years of age and older
* Provided informed consent to participate in the registry
* English speaking
* Agrees to complete a survey at specified time points from baseline to 12 Months

Exclusion Criteria:

* Physician discretion
* Vulnerable populations

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Premenopausal women with heavy menstrual bleeding due to benign causes for whom child bearing is complete.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Re-intervention rate | 12 Months
  The cumulative re-intervention rate at 12 months will be compared to the pivotal clinical study.
Site of service rate | 12 Months
  The mix of Cerene treatments performed at different sites of service will be tabulated.
Patient quality of life | 12 Months
  The patient's quality of life at baseline and 12 Months will be compared.

SECONDARY OUTCOMES:
Physician survey | 12 Months
  Each physician user will be surveyed on several topics related to the device.
Cost analysis | 12 Months
  A cost analysis of Cerene treatments for different sites of service may be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Yu, MBA, Study Chair — Executive VP of Regulatory, Clinical, and Medical Affairs
Locations (2):
- United States (2):
  - Axia Women's Health / Rubino OB/GYN Group, West Orange, New Jersey
  - Seven Hills Women's Health Centers, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Curlin HL, Cintron LC, Anderson TL. A Prospective, Multicenter, Clinical Trial Evaluating the Safety and Effectiveness of the Cerene Device to Treat Heavy Menstrual Bleeding. J Minim Invasive Gynecol. 2021 Apr;28(4):899-908. doi: 10.1016/j.jmig.2020.08.013. Epub 2020 Aug 22. PMID 32835865